CLINICAL TRIAL: NCT00048061
Title: Randomized, Double-blind, Double Dummy, Parallel Groups, Multicenter Study to Compare the Efficacy and Safety of Monthly Oral Administration of 100 mg and 150 mg Ibandronate With 2.5 mg Daily Oral Ibandronate in Postmenopausal Osteoporosis
Brief Title: MOBILE Study - A Study of Bonviva (Ibandronate) Regimens in Women With Post-Menopausal Osteoporosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BM16549
Record Dates: First submitted 2002-10-24; First posted 2002-10-25 (Estimated); Results first posted 2016-05-30 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2018-02

CONDITIONS: Post Menopausal Osteoporosis
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Ibandronic Acid; Calcium; Vitamin D

ARMS (4):
- Ibandronate 2.5 mg (Active Comparator): Participants will receive 2.5 milligram (mg) ibandronate Per oral (PO) daily and an oblong placebo tablet PO monthly. Participants will also receive calcium 500 mg /day and vitamin D 400 international units (IU)/day .
  Interventions: Drug: Ibandronate [Bonviva/Boniva]; Dietary Supplement: Calcium; Dietary Supplement: Vitamin D
- Ibandronate 50/50 mg (Experimental): Participants will receive 100 mg ibandronate PO monthly taken on a single day (2 X 50 mg tablets) and round placebo tablet PO daily. Participants will also receive calcium 500 mg /day and vitamin D 400 IU/day.
  Interventions: Drug: Ibandronate [Bonviva/Boniva]; Dietary Supplement: Calcium; Dietary Supplement: Vitamin D
- Ibandronate 100 mg (Experimental): Participants will receive 100 mg ibandronate PO monthly divided over two consecutive days (50 mg tablet/day) and a round placebo tablet PO daily. Participants will also receive calcium 500 mg /day and vitamin D 400 IU/day
  Interventions: Drug: Ibandronate [Bonviva/Boniva]; Dietary Supplement: Calcium; Dietary Supplement: Vitamin D
- Ibandronate 150 mg (Experimental): Participants will receive 150 mg ibandronate PO monthly taken on a single day and a round placebo tablet PO daily. Participants will also receive calcium 500 mg /day and vitamin D 400 IU/day
  Interventions: Drug: Ibandronate [Bonviva/Boniva]; Dietary Supplement: Calcium; Dietary Supplement: Vitamin D

INTERVENTIONS:
Drug: Ibandronate [Bonviva/Boniva] — 2.5mg po daily
  Arms: Ibandronate 2.5 mg
Drug: Ibandronate [Bonviva/Boniva] — 100mg po monthly on a single day
  Arms: Ibandronate 50/50 mg
Drug: Ibandronate [Bonviva/Boniva] — 100mg po monthly over 2 consecutive days
  Arms: Ibandronate 100 mg
Drug: Ibandronate [Bonviva/Boniva] — 150mg po monthly
  Arms: Ibandronate 150 mg
Dietary Supplement: Calcium — 500 mg/day
Dietary Supplement: Vitamin D — 400 IU/day

SUMMARY:
This study will compare the efficacy and safety of different treatment regimens of oral Bonviva tablets in women with post-menopausal osteoporosis. Patients will also receive daily supplementation with vitamin D and calcium. The anticipated time of study treatment is 2+ years, and the target sample size is 500+ individuals.

ELIGIBILITY:
Inclusion Criteria:

* women 55-80 years of age;
* post-menopausal for >= 5 years;
* ambulatory.

Exclusion Criteria:

* malignant disease diagnosed within the previous 10 years (except basal cell cancer that has been successfully removed);
* breast cancer within the previous 20 years;
* allergy to bisphosphonates;
* previous treatment with an intravenous bisphosphonate at any time;
* previous treatment with an oral bisphosphonate within the last 6 months, >1 month of treatment within the last year, or >3 months of treatment within the last 2 years.

Ages: 55 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1609 (Actual)
Dates: Start 2002-04; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (65):
- United States (20):
  - Irvine, California
  - Loma Linda, California
  - Los Angeles, California
  - Oakland, California
  - Rancho Mirage, California
  - Lakewood, Colorado
  - Gainesville, Florida
  - Bethesda, Maryland
  - Wheaton, Maryland
  - St Louis, Missouri
  - Billings, Montana
  - Omaha, Nebraska
  - Livingston, New Jersey
  - Albuquerque, New Mexico
  - Portland, Oregon
  - Wyomissing, Pennsylvania
  - San Antonio, Texas
  - Richmond, Virginia
  - Seattle, Washington
  - Madison, Wisconsin
- Australia (3):
  - Adelaide
  - Parkville
  - Perth
- Belgium (2):
  - Liège
  - Merksem
- Brazil (4):
  - Campinas
  - Curitiba
  - Porto Alegre
  - São Paulo
- Canada (4):
  - Calgary, Alberta
  - Vancouver, British Columbia
  - Toronto, Ontario
  - Québec, Quebec
- Czechia (2):
  - Pilsen
  - Prague
- Denmark (3):
  - Aalborg
  - Ballerup Municipality
  - Vejle
- France (2):
  - Caen
  - Lyon
- Germany (2):
  - Berlin
  - Hanover
- Hungary (4):
  - Balatonfüred
  - Budapest
  - Kiskunhalas
  - Zalaegerszeg
- Italy (2):
  - Siena
  - Valeggio sul Mincio
- Mexico (2):
  - León
  - Obregón
- Norway (3):
  - Haugesund
  - Oslo
  - Stavanger
- Poland (2):
  - Krakow
  - Warsaw
- Bucharest, Romania
- South Africa (2):
  - Cape Town
  - Johannesburg
- Spain (2):
  - Barcelona
  - Madrid
- Zurich, Switzerland
- United Kingdom (4):
  - Cardiff
  - Liverpool
  - London
  - Southampton

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted from 26 April 2002 to 08 Dec 2004 across 65 centers in the world.
Pre-assignment Details: A total of 1609 participants were randomized, of which 1602 received the study drug.
Groups:
- Ibandronate 2.5 mg: Participants received 2.5 milligram (mg) ibandronate Per oral (PO) daily and an oblong placebo tablet PO monthly Participants also received calcium 500 mg /day and vitamin D 400 international units (IU) per day.
- Ibandronate 50/50 mg: Participants received 100 mg ibandronate PO monthly taken on a single day (2 X 50 mg tablets) and round placebo tablet PO daily. Participants also received calcium 500 mg /day and vitamin D 400 IU/day.
- Ibandronate 100 mg: Participants received 100 mg ibandronate PO monthly divided over two consecutive days (50 mg tablet/day) and a round placebo tablet PO daily. Participants also received calcium 500 mg /day and vitamin D 400 IU/day.
- Ibandronate 150 mg: Participants received 150 mg ibandronate PO monthly taken on a single day and a round placebo tablet PO daily. Participants also received calcium 500 mg /day and vitamin D 400 IU/day.
Period: Overall Study
Arm/Group | Ibandronate 2.5 mg | Ibandronate 50/50 mg | Ibandronate 100 mg | Ibandronate 150 mg
Started | 400 | 401 | 400 | 401
Completed | 325 | 328 | 316 | 322
Not Completed | 75 | 73 | 84 | 79
Not completed — Adverse Event | 41 | 32 | 44 | 37
Not completed — Lost to Follow-up | 3 | 2 | 4 | 5
Not completed — Withdrawal by Subject | 20 | 29 | 29 | 32
Not completed — Did not follow-up | 5 | 5 | 4 | 5
Not completed — Early improvement | 6 | 5 | 3 | 0

BASELINE CHARACTERISTICS:
Population: The safety population consisted of all participants who were randomized and received at least one dose of the study medication, and who have at least one follow-up data point.
Groups:
- Ibandronate 2.5 mg: Participants received 2.5 mg ibandronate PO daily and an oblong placebo tablet PO monthly Participants also received calcium 500 mg /day and vitamin D 400 IU/day.
- Total: Total of all reporting groups
Arm/Group | Ibandronate 2.5 mg | Ibandronate 50/50 mg | Ibandronate 100 mg | Ibandronate 150 mg | Total
Number analyzed (Participants) | 395 | 396 | 396 | 396 | 1583
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.8 (6.61) | 66.0 (6.71) | 66.2 (6.38) | 66.2 (6.64) | 66.0 (6.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 395 | 396 | 396 | 396 | 1583
  Male | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Relative Change From Baseline at One Year (12 Months) in Mean Lumbar Spine (L2 - L4) Bone Mineral Density
Description: Relative change in Bone Mineral Density (BMD) is the percentage change from baseline of BMD of vertebrae L2 - L4 that are not fractured and not affected by an osteoarthritic process to such a degree that accurate measurement of BMD would be considered jeopardized by the central reading center after 12 months of treatment. It is calculated as the sum of bone mineral content divided by the sum of area of all lumbar vertebrae L2 - L4 that are not fractured and not affected by an osteoarthritic process at Month 12. Participants available at particular time point for assessment were included in the analysis.
Time Frame: From Baseline (Month 0) to Month 12
Population: The per-protocol(PP) population included participants in Intent-to-treat(ITT) population who were randomized, received at least one dose of medication and had at least one valid efficacy(BMD or Serum CTX)follow-up data point;defined as any measurement that can be scientifically compared to baseline measurement, and had no major protocol violations.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Ibandronate 2.5 mg | Ibandronate 50/50 mg | Ibandronate 100 mg | Ibandronate 150 mg
Number analyzed (Participants) | 314 | 322 | 306 | 314
Percent change | 3.7427 (4.0149) | 4.3395 (3.9557) | 4.0328 (3.6815) | 4.7611 (3.8931)
Statistical Analysis 1: Comparison: Ibandronate 2.5 mg vs Ibandronate 50/50 mg; Test type: Non-Inferiority or Equivalence — The monthly dosing regimen (Ibandronate 50/50 mg monthly) was considered non-inferior to the 2.5 mg daily regimen if the lower bound of the two-sided 95% CI on the difference in mean percent change in BMD was greater or equal to -1 percentage point; p = 0.045, ANOVA; Mean Difference (Final Values) = 0.615, 95% CI 2-sided [0.013 to 1.216] — Treatment effect is the difference in the mean values of the monthly oral dose regimens (Ibandronate 50/50) and the active-control
Statistical Analysis 2: Comparison: Ibandronate 2.5 mg vs Ibandronate 100 mg; Test type: Non-Inferiority or Equivalence — The monthly dosing regimen (Ibandronate 100 mg) was considered non-inferior to the 2.5 mg daily regimen if the lower bound of the two-sided 95% CI on the difference in mean percent change in BMD was greater or equal to -1 percentage point; p = 0.338, ANOVA; Mean Difference (Final Values) = 0.297, 95% CI 2-sided [-0.312 to 0.906] — Treatment effect is the difference in the mean values of the monthly oral dose regimens (Ibandronate 100 mg) and the active-control
Statistical Analysis 3: Comparison: Ibandronate 2.5 mg vs Ibandronate 150 mg; Test type: Non-Inferiority or Equivalence — The monthly dosing regimen (Ibandronate 150 mg) was considered non-inferior to the 2.5 mg daily regimen if the lower bound of the two-sided 95% CI on the difference in mean percent change in BMD was greater or equal to -1 percentage point; p = 0.001, ANOVA; Mean Difference (Final Values) = 1.000, 95% CI 2-sided [0.395 to 1.605] — Treatment effect is the difference in the mean values of the monthly oral dose regimens (Ibandronate 150 mg) and the active-control

2. Secondary Outcome: Relative Change From Baseline at Two Years (24 Months) in Mean Lumbar Spine (L2-L4) BMD
Description: Relative change in BMD is the percentage change from baseline of BMD of vertebrae L2 - L4 that are not fractured and not affected by an osteoarthritic process to such a degree that accurate measurement of BMD would be considered jeopardized by the central reading center after 24 months of treatment. It is calculated as the sum of bone mineral content divided by the sum of area of all lumbar vertebrae L2 - L4 that are not fractured and not affected by an osteoarthritic process at Month 24.
Time Frame: From Baseline (Month 0) to Month 24
Population: The PP population consisted of all participants in the ITT population who had no major violations of the protocol.Participants available at particular time point for assessment were included in the analysis.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Ibandronate 2.5 mg | Ibandronate 50/50 mg | Ibandronate 100 mg | Ibandronate 150 mg
Number analyzed (Participants) | 294 | 294 | 278 | 291
Percent change | 4.9623 (4.6525) | 5.3350 (4.8235) | 5.5760 (4.2280) | 6.5503 (4.5118)

3. Secondary Outcome: Absolute Change From Baseline at One Year (12 Months) and Two Years (24 Months) in Mean Lumbar Spine (L2-L4) BMD
Description: The absolute change (g/cm^2) from baseline in mean BMD of the lumbar spine (L2 - L4) at one and two years. A difference in the mean values between the active groups and the control was calculated.
Time Frame: From Baseline (Month 0) to Months 12 and 24
Population: The PP population consisted of all participants in the ITT population who had no major violations of the protocol. n = number of participants evaluable at particular time of assessment.
Measure: Mean (Standard Deviation); unit: g/cm2
Arm/Group | Ibandronate 2.5 mg | Ibandronate 50/50 mg | Ibandronate 100 mg | Ibandronate 150 mg
Number analyzed (Participants) | 314 | 322 | 306 | 314
g/cm2
  At 12 months, n = 314, 322, 306, 314 | 0.028 (0.0291) | 0.033 (0.0298) | 0.030 (0.0271) | 0.036 (0.0290)
  At 24 months, n = 294, 294, 278, 291 | 0.036 (0.0337) | 0.039 (0.0355) | 0.042 (0.0313) | 0.049 (0.0330)

4. Secondary Outcome: Relative Change From Baseline at One Year (12 Months) and Two Years (24 Months) in Mean Proximal Femur ( Total Hip, Trochanter, Femoral Neck) BMD
Description: Proximal femur BMD was measured by dual-energy X ray absorptiometry at baseline, after one and two years of treatment and was read by a central reading center.
Time Frame: From Baseline (Month 0) to Months 12 and 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Ibandronate 2.5 mg | Ibandronate 50/50 mg | Ibandronate 100 mg | Ibandronate 150 mg
Number analyzed (Participants) | 315 | 319 | 306 | 316
Percent change
  Total hip At Month 12, n = 315,319,306,316 | 1.9626 (2.8311) | 2.2172 (2.7504) | 2.6878 (2.6646) | 3.0092 (2.7105)
  Total hip At Month 24, n = 292,291,277,289 | 2.4955 (3.0884) | 2.8132 (3.2408) | 3.5165 (3.2831) | 4.1601 (2.8335)
  Trochanter At Month 12, n = 315,319,306,316 | 3.1917 (4.1268) | 3.4931 (4.0876) | 3.8226 (3.7077) | 4.5904 (3.9436)
  Trochanter At Month 24, n = 292,291,277,289 | 4.0204 (4.3460) | 4.6289 (4.5518) | 5.3135 (4.7335) | 6.1755 (4.2550)
  Femoral neck At Month 12, n = 315,319,306,316 | 1.7164 (3.6233) | 1.8141 (3.4391) | 1.8797 (3.4998) | 2.1914 (3.4842)
  Femoral neck At Month 24, n=292,291,277,289 | 1.9087 (4.2212) | 2.0581 (4.1189) | 2.6209 (3.8339) | 3.1195 (4.0549)

5. Secondary Outcome: Absolute Change From Baseline at One Year (12 Months) and Two Years (24 Months) in Mean Proximal Femur ( Total Hip, Trochanter, Femoral Neck) BMD.
Description: Proximal femur BMD was measured by dual-energy X-ray absorptiometry at baseline, after one and two years of treatment and was read by a central reading center
Time Frame: From Baseline (Month 0) to Months 12 and 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: g/cm2
Arm/Group | Ibandronate 2.5 mg | Ibandronate 50/50 mg | Ibandronate 100 mg | Ibandronate 150 mg
Number analyzed (Participants) | 315 | 319 | 306 | 316
g/cm2
  Total hip At Month 12, n = 315,319,306,316 | 0.014 (0.0204) | 0.016 (0.0205) | 0.020 (0.0190) | 0.022 (0.0190)
  Total hip At Month 24, n = 292,291,277,290 | 0.018 (0.0225) | 0.021 (0.0241) | 0.026 (0.0237) | 0.031 (0.0199)
  Trochanter At Month 12, n = 315,319,306,316 | 0.018 (0.0228) | 0.020 (0.0238) | 0.022 (0.0206) | 0.026 (0.0211)
  Trochanter At Month 24, n = 292,291,277,290 | 0.023 (0.0241) | 0.027 (0.0259) | 0.030 (0.0263) | 0.035 (0.0231)
  Femoral neck At Month 12, n = 315,319,306,316 | 0.011 (0.0230) | 0.011 (0.0226) | 0.012 (0.0228) | 0.014 (0.0224)
  Femoral neck At Month 24, n = 315,319,306,316 | 0.012 (0.0265) | 0.013 (0.0272) | 0.017 (0.0248) | 0.020 (0.0257)

6. Secondary Outcome: Percentage of Participants With Mean Lumbar Spine (L2 - L4) BMD Above or Equal to Baseline at Months 12 and 24
Description: A participant is a responder if the mean lumber spine (L2 - L4) BMD had remained the same or increased above baseline.
Time Frame: Months 12 and 24
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Ibandronate 2.5 mg | Ibandronate 50/50 mg | Ibandronate 100 mg | Ibandronate 150 mg
Number analyzed (Participants) | 314 | 322 | 306 | 314
Percentage of participants
  At Month 12, n = 314,322,306,314 | 83.8 | 87.6 | 86.6 | 90.8
  At Month 24, n = 294,294,278,291 | 86.4 | 87.8 | 87.8 | 93.5

7. Secondary Outcome: Percentage of Participants With Total Hip BMD Above or Equal to Baseline at Months 12 and 24
Description: A participant is a responder if the mean total hip BMD had remained the same or increased above baseline.
Time Frame: Months 12 and 24
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Ibandronate 2.5 mg | Ibandronate 50/50 mg | Ibandronate 100 mg | Ibandronate 150 mg
Number analyzed (Participants) | 315 | 319 | 306 | 306
Percentage of participants
  At Month 12, n = 315,319,306,306 | 76.8 | 81.2 | 86.9 | 90.5
  At Month 24, n = 292,291,277,289 | 78.4 | 83.2 | 88.8 | 93.4

8. Secondary Outcome: Percentage of Participants With Trochanter BMD Above or Equal to Baseline at Months 12 and 24
Description: A participant is a responder if the mean trochanter BMD had remained the same or increased above baseline.
Time Frame: Months 12 and 24
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Ibandronate 2.5 mg | Ibandronate 50/50 mg | Ibandronate 100 mg | Ibandronate 150 mg
Number analyzed (Participants) | 315 | 319 | 306 | 316
Percentage of participants
  At Month 12, n = 315,319,306,316 | 80.0 | 83.1 | 88.2 | 92.4
  At Month 24, n = 292,291,277,289 | 84.2 | 86.6 | 89.9 | 94.1

9. Secondary Outcome: Percentage of Participants With Femoral Neck BMD Above or Equal to Baseline at Months 12 and 24
Description: A participant is a responder if the mean femoral neck BMD had remained the same or increased above baseline.
Time Frame: Months 12 and 24
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Ibandronate 2.5 mg | Ibandronate 50/50 mg | Ibandronate 100 mg | Ibandronate 150 mg
Number analyzed (Participants) | 315 | 319 | 306 | 316
Percentage of participants
  At Month 12, n = 315,319,306,316 | 71.1 | 72.4 | 69.0 | 75.3
  At Month 24, n = 292,291,277,289 | 69.2 | 71.1 | 78.7 | 81.0

10. Secondary Outcome: Percentage of Participants With Mean Total Hip and Lumbar Spine BMD Above or Equal to Baseline at Months 12 and 24
Description: A participant is a responder if the mean total hip and mean lumbar spine BMD had remained the same or increased above baseline.
Time Frame: Months 12 and 24
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Ibandronate 2.5 mg | Ibandronate 50/50 mg | Ibandronate 100 mg | Ibandronate 150 mg
Number analyzed (Participants) | 314 | 318 | 304 | 310
Percentage of participants
  At Month 12, n = 314,318,304,310 | 65.6 | 72.3 | 77.6 | 83.5
  At Month 24, n = 292,291,276,287 | 70.5 | 75.3 | 79.3 | 87.1

11. Secondary Outcome: Percentage of Participants With Mean Trochanter and Lumbar Spine BMD Above or Equal to Baseline at Months 12 and 24
Description: A participant is a responder if the mean trochanter and lumbar spine BMD had remained the same or increased above baseline.
Time Frame: Months 12 and 24
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Ibandronate 2.5 mg | Ibandronate 50/50 mg | Ibandronate 100 mg | Ibandronate 150 mg
Number analyzed (Participants) | 314 | 318 | 304 | 310
Percentage of participants
  At Month 12, n = 314,318,304,310 | 68.8 | 75.5 | 78.0 | 84.2
  At Month 24, n = 292,291,276,287 | 75.7 | 77.3 | 80.1 | 88.2

12. Secondary Outcome: Percentage of Participants With Mean Femoral Neck and Lumbar Spine BMD Above or Equal to Baseline at Months 12 and 24
Description: A participant is a responder if the mean femoral neck and lumbar spine BMD had remained the same or increased above baseline.
Time Frame: Months 12 and 24
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Ibandronate 2.5 mg | Ibandronate 50/50 mg | Ibandronate 100 mg | Ibandronate 150 mg
Number analyzed (Participants) | 314 | 318 | 304 | 310
Percentage of participants
  At Month 12, n = 314,318,304,310 | 62.4 | 64.5 | 60.9 | 68.7
  At Month 24, n = 292,291,276,287 | 63.4 | 63.9 | 71.0 | 75.6

13. Secondary Outcome: Relative Change In Baseline in Serum C-telopeptide of Alpha-chain of Type I Collagen [ CTX] ] to Months 3, 6, 12, and 24
Description: Serum CTX, a biochemical marker of bone resorption, was assessed using the Elecsys S-CTX-I assay (an ElectroChemiLuminescence Immunoassay (ECLIA) Technique).
Time Frame: From Baseline (Month 0) to Months 3, 6, 12, 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Ibandronate 2.5 mg | Ibandronate 50/50 mg | Ibandronate 100 mg | Ibandronate 150 mg
Number analyzed (Participants) | 272 | 278 | 276 | 278
Percent change
  At Month 3, n = 269,278,271,276 | -49.5458 (30.8286) | -46.4771 (26.5096) | -50.2368 (28.1576) | -57.3433 (33.9505)
  At Month 6, n = 270,272,274,278 | 55.5900 (34.1672) | -53.9838 (27.3557) | -55.9614 (31.2801) | -66.4354 (25.4762)
  At Month 12, n = 272,276,276,267 | -58.8244 (29.8250) | -57.5363 (27.2271) | -58.1046 (33.5095) | -67.0703 (41.4563)
  At Month 24, n = 221,215,211,235 | -51.2360 (37.9032) | -51.3040 (27.9844) | -49.5567 (44.9707) | 61.8822 (28.2309)

14. Secondary Outcome: Absolute Change In Baseline in Serum CTX to Months 12 and 24
Description: as for outcome 13
Time Frame: From Baseline (Month 0) to Months 12 and 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Ibandronate 2.5 mg | Ibandronate 50/50 mg | Ibandronate 100 mg | Ibandronate 150 mg
Number analyzed (Participants) | 272 | 276 | 276 | 267
ng/ml
  Month 12, n = 272, 276, 276, 267 | -0.323 (0.2292) | -0.326 (0.2212) | -0.340 (0.2287) | -0.377 (0.2135)
  Month 24, n = 221, 215, 211, 235 | -0.285 (0.2052) | -0.298 (0.1980) | -0.312 (0.2398) | -0.340 (0.2062)

15. Secondary Outcome: Number of Participants With Any Adverse Events and Serious Adverse Event
Description: An Adverse Event (AE) is any untoward medical occurrence in a participant or clinical investigation subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. A serious adverse event (SAE) is any untoward medical occurrence that at any dose results in death, are life threatening, requires hospitalization or prolongation of hospitalization or results in disability/incapacity, and congenital anomaly/birth defect.
Time Frame: Up to Month 24
Population: as for baseline characteristics
Measure: Number; unit: Participants
Arm/Group | Ibandronate 2.5 mg | Ibandronate 50/50 mg | Ibandronate 100 mg | Ibandronate 150 mg
Number analyzed (Participants) | 395 | 396 | 396 | 396
Participants
  Any AE | 302 | 313 | 318 | 317
  SAE | 38 | 54 | 55 | 45

16. Secondary Outcome: Number Of Participants With Marked Laboratory Abnormalities
Description: Marked laboratory abnormalities were defined as those values that were outside the reference range and showed a clinically relevant change from baseline. The reference range for hemoglobin was 110-200 (gram per liter [g/L]), hematocrit was 0.31-0.56 fraction, white blood cells (WBC) was 3.0-18.0 (10*9/L), serum glutamic-pyruvic transaminase (SGPT/ALT) was 0-110 IU/L, blood urea nitrogen (BUN) was 0.0-14.3 (millimoles per Liter [mmol/L]), Chloride was 95-115 (mmol/L), Potassium was 3.0 - 6.0 (mmol/L), Sodium was 130-150 (mmol/L), Calcium was 2.00-2.90 (mmol/L), Phosphate was 0.75 - 1.60 (mmol/L) and Creatinine was 0- 154 (micromoles/liter [umol/L].
Time Frame: Up to Month 24
Population: The safety population consisted of all participants who were randomized and received at least one dose of the study medication, and who have at least one follow-up data point. n = number of participants evaluable at particular time of assessment.
Measure: Number; unit: Participants
Arm/Group | Ibandronate 2.5 mg | Ibandronate 50/50 mg | Ibandronate 100 mg | Ibandronate 150 mg
Number analyzed (Participants) | 390 | 390 | 385 | 385
Participants
  Hematocrit Low, n = 389,387,382,385 | 2 | 0 | 1 | 3
  Hemoglobin High, n = 389,389,382,385 | 0 | 0 | 1 | 0
  Hemoglobin Low, n = 389,389,382,385 | 3 | 3 | 6 | 3
  WBC Low, n = 389,389,382,385 | 1 | 1 | 4 | 4
  ALT (SGPT) High, n = 390,390,385,385 | 9 | 8 | 8 | 8
  BUN High, n = 390,390,385,385 | 2 | 0 | 0 | 0
  Creatinine High, n = 390,390,385,385 | 1 | 1 | 0 | 1
  Chloride Low, n =3 89,390,385,384 | 3 | 3 | 0 | 3
  Potassium Low, n = 389,390,385,383 | 0 | 0 | 0 | 1
  Sodium High, n = 389,390,385,384 | 0 | 0 | 1 | 2
  Sodium Low, n = 389,390,385,384 | 2 | 1 | 0 | 0
  Calcium High, n = 390,390,385,385 | 1 | 0 | 0 | 1
  Phosphate High, n = 390,390,385,385 | 4 | 3 | 3 | 1
  Phosphate Low, n = 390,390,385,385 | 2 | 2 | 2 | 1

ADVERSE EVENTS:
Time Frame: 24 months
Description: SAEs and non-serious AEs were reported for members of the Safety Population, comprised of participants who were randomized and had at least one dose of study drug, whether withdrawn prematurely or not, and who had at least one follow-up data point.
Arm/Group | Ibandronate 2.5 mg | Ibandronate 50/50 mg | Ibandronate 100 mg | Ibandronate 150 mg
Serious Adverse Events (participants affected / at risk) | 38/395 | 54/396 | 55/396 | 45/396
Other Adverse Events (participants affected / at risk) | 190/395 | 190/396 | 191/396 | 182/396
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ibandronate 2.5 mg (N=395) | Ibandronate 50/50 mg (N=396) | Ibandronate 100 mg (N=396) | Ibandronate 150 mg (N=396)
Pneumonia (Infections and infestations) | 3 | 1 | 2 | 2
Cellulitis (Infections and infestations) | 1 | 1 | 0 | 0
Lower respiratory tract Infection (Infections and infestations) | 0 | 0 | 1 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 1
Bronchial infection (Infections and infestations) | 0 | 0 | 1 | 0
Chronic sinusitis (Infections and infestations) | 1 | 0 | 0 | 0
Conjunctivitis bacterial (Infections and infestations) | 1 | 0 | 0 | 0
Dacryocystitis infective (Infections and infestations) | 1 | 0 | 0 | 0
Ear infection (Infections and infestations) | 0 | 0 | 0 | 1
Ear infection viral (Infections and infestations) | 0 | 0 | 1 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 1
Gangrene (Infections and infestations) | 0 | 0 | 1 | 0
Hematoma infection (Infections and infestations) | 0 | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 0 | 0
Laryngopharyngitis (Infections and infestations) | 0 | 0 | 1 | 0
Postoperative abscess (Infections and infestations) | 1 | 0 | 0 | 0
Pulmonary tuberculosis (Infections and infestations) | 1 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 1
Salmonellosis (Infections and infestations) | 0 | 0 | 0 | 1
Superinfection (Infections and infestations) | 0 | 0 | 1 | 0
Superinfection lung (Infections and infestations) | 0 | 0 | 1 | 0
Urosepsis (Infections and infestations) | 1 | 0 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 1 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 1 | 1
Melaena (Gastrointestinal disorders) | 2 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Colonic polyp (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Gastrointestinal haemorrhage (Infections and infestations) | 0 | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Appendicitis perforated (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Colitis ulcerative (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Erosive duodenitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Reflux gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 0 | 3
Myocardial ischemia (Cardiac disorders) | 1 | 1 | 0 | 2
Acute myocardial infarction (Cardiac disorders) | 2 | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 1 | 1 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 2 | 0 | 0
Coronary artery disease (Cardiac disorders) | 1 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 2 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 1 | 0 | 0
Angina unstable (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 0 | 0 | 1 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 1 | 0 | 0
Left ventricular failure (Cardiac disorders) | 0 | 1 | 0 | 0
Tachyarrhythmia (Cardiac disorders) | 1 | 0 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 1
Cardiac pacemaker malfunction (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Meniscus lesion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Pain trauma activated (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Patella fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Pubic rami fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Vascular graft occlusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Benign neoplasm of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Gammopathy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Ovarian epithelial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 2 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 1 | 0
Vertebrobasilar insufficiency (Nervous system disorders) | 0 | 1 | 0 | 1
Aphasia (Nervous system disorders) | 0 | 0 | 1 | 0
Dementia alzheimer's type (Nervous system disorders) | 0 | 0 | 1 | 0
Embolic stroke (Nervous system disorders) | 1 | 0 | 0 | 0
Facial palsy (Nervous system disorders) | 0 | 0 | 1 | 0
Facial paresis (Nervous system disorders) | 0 | 0 | 1 | 0
Haemorrhagic cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 1
Loss of consciousness (Nervous system disorders) | 1 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 1
Parkinson's disease (Nervous system disorders) | 0 | 1 | 0 | 0
Parkinsonism (Nervous system disorders) | 0 | 0 | 1 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 1 | 0
Localised osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 4 | 1 | 2
Back pain (Nervous system disorders) | 1 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Osteitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Spondylosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Toe deformity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 2 | 0 | 1
Aortic aneurysm (Vascular disorders) | 0 | 1 | 0 | 1
Haematoma (Vascular disorders) | 0 | 1 | 1 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0
Intermittent claudication (Vascular disorders) | 0 | 0 | 0 | 1
Vascular pseudoaneurysm (Vascular disorders) | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 | 2 | 2 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0
Bipolar disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Major depression (Psychiatric disorders) | 0 | 0 | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Chronic obstructive airways disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Laryngeal polyp (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 1 | 1
Cystocele (Renal and urinary disorders) | 0 | 0 | 1 | 0
Renal colic (Renal and urinary disorders) | 0 | 0 | 0 | 1
Urethral syndrome (Renal and urinary disorders) | 0 | 0 | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0 | 0
Cervical polyp (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Endometrial hypertrophy (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Pelvic prolapse (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Uterine prolapse (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Vaginal prolapse (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Autoimmune thyroiditis (Endocrine disorders) | 0 | 0 | 0 | 1
Hyperparathyroidism (Endocrine disorders) | 0 | 0 | 1 | 0
Hyperparathyroidism primary (Endocrine disorders) | 0 | 0 | 0 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 2
Adverse drug reaction (General disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 1 | 0
Bile duct obstruction (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Liver disorder (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Cataract (Eye disorders) | 0 | 1 | 0 | 0
Diplopia (Eye disorders) | 0 | 1 | 0 | 0
Macular hole (Eye disorders) | 0 | 0 | 0 | 1
Cutaneous lupus erythematosus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin necrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Cyst removal (Surgical and medical procedures) | 0 | 1 | 0 | 0
Eventration procedure (Surgical and medical procedures) | 1 | 0 | 0 | 0
Dermoid cyst of ovary (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0
Vestibular neuronitis (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ibandronate 2.5 mg (N=395) | Ibandronate 50/50 mg (N=396) | Ibandronate 100 mg (N=396) | Ibandronate 150 mg (N=396)
Arthralgia (Musculoskeletal and connective tissue disorders) | 24 | 39 | 35 | 27
Back pain (Musculoskeletal and connective tissue disorders) | 25 | 36 | 36 | 28
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 | 14 | 13 | 20
Localised osteoarthritis (Musculoskeletal and connective tissue disorders) | 10 | 12 | 12 | 19
Nasopharyngitis (Infections and infestations) | 38 | 23 | 27 | 24
Influenza (Infections and infestations) | 25 | 31 | 18 | 26
Urinary tract infection (Infections and infestations) | 15 | 18 | 15 | 19
Bronchitis (Infections and infestations) | 20 | 10 | 18 | 12
Nausea (Gastrointestinal disorders) | 20 | 19 | 18 | 25
Diarrhoea (Gastrointestinal disorders) | 21 | 20 | 16 | 19
Dyspepsia (Gastrointestinal disorders) | 28 | 29 | 37 | 26
Hypertension (Vascular disorders) | 46 | 43 | 47 | 41
Hypercholesterolaemia (Metabolism and nutrition disorders) | 21 | 9 | 16 | 18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights